CLINICAL TRIAL: NCT05638009
Title: The ECLA/PHRI Intervention in the Community Trial - EPIC Trial
Brief Title: The ECLA/PHRI Intervention in the Community Trial
Acronym: EPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Estudios Clínicos Latino América (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EPIC. Version 2.0
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Hypertension
Keywords: Sodium Chloride; Dietary
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): regular salt (99% sodium chloride)
- Salt substitute 1 (Experimental): Salt substitute 1 is a potassium-enriched salt substitute composed of 66% potassium chloride and 33% sodium chloride
  Interventions: Dietary Supplement: Salt substitute 66%33%
- Salt substitute 2 (Experimental): Salt substitute 2 is a potassium-enriched salt substitute composed of 33% potassium chloride and 66% sodium chloride
  Interventions: Dietary Supplement: Salt substitute 33%/66%

INTERVENTIONS:
Dietary Supplement: Salt substitute 66%33% — Salt substitute composed of 66% potassium chloride and 33% sodium chloride
  Arms: Salt substitute 1
Dietary Supplement: Salt substitute 33%/66% — Salt substitute composed of 33% potassium chloride and 66% sodium chloride
  Arms: Salt substitute 2

SUMMARY:
EPIC is a cluster-randomized, double-blind trial to evaluate the effect of two potassium-enriched salt substitute preparations (one available in the Argentine market and one derived from it), compared to regular salt on systolic blood pressure in subjects ≥ 18 and ≤ 90 years old from Rosario department households in Santa Fe Province, Argentina.

DETAILED DESCRIPTION:
The effect of reduced sodium salt preparations has been evaluated in clinical studies (observational and randomized clinical trials) and in meta-analyses, and although a reduction in blood pressure was observed, they have particular characteristics that make them difficult to extrapolate their results to Western populations.

In one of these trials, conducted in rural Indian hypertensive patients, the use of a salt substitute of 75% sodium chloride and 25% potassium chloride showed a significant reduction of systolic blood pressure with a mean difference of -4.58 mmHg in 3 months from baseline to the end of the trial.

Recently, a large cluster-randomized trial conducted in 600 villages in rural areas of five provinces of China (SSaSS trial) among patients with a history of stroke or 60 years of age or elder with elevated blood pressure showed that stroke rates, major cardiovascular events and death from any cause were significantly lower with a salt substitute than with regular salt. The salt substitute used in this trial had 1/3 less sodium than regular salt and substantially more potassium. Therefore, the salt substitute led to an 8% less sodium intake but a 50% higher intake in potassium. This suggests that the greatest impact of salt substitution in this RCT may have been due to an increase in potassium intake rather than the modest decrease in sodium intake that was associated with an average reduction of 2.65 mmHg for SBP (-4.32 to -0.97) and +0.30 mmHg (-0.72 to +1.32) for DBP. In addition, the mean sodium intake in the studied population in this trial was approximately 4.2 gr/d, which is higher than the global average worldwide sodium consumption of 3.9 gr/d. In contrast, potassium intake was lower than the average global potassium intake. Therefore, several considerations that limit the applicability to other populations remain unresolved. The sodium intake of the Chinese rural population is higher than in many other countries, while the potassium intake is relatively low. In addition, in many countries commercially available foods may have added sodium chloride for preservation and thus increase the amount of sodium to the diet. Therefore, the use of salt substitutes would not fully account for salt intake in most cases. Finally, Chinese social and environmental features may be somewhat different to most western countries.

EPIC's investigators stated the hypothesis that salt substitutes could lower systolic blood pressure in a dose-response mode. Therefore, they propose to conduct a randomized cluster trial to evaluate the effect of consuming two doses enriched potassium salt substitutes preparations compared to regular salt intake on systolic blood pressure in individuals from Rosario department.

ELIGIBILITY:
Inclusion Criteria:

Subjects ≥ 18 and ≤ 90 years old will be included, with no specific clinical conditions from households that meets the following criteria:

* The household must be composed of at least 2 individuals
* At least 1 of the individuals included must be over 40 years of age
* The household must be located in Rosario department, Santa Fe province, Argentina

Exclusion Criteria:

Households will be excluded if a any household member has a at least one of the following contraindication to the salt substitute used in the trial:

* use of a potassium-sparing diuretic
* use of a potassium supplement
* known history of hyperkalemia
* use of salt reduced in sodium and enriched in potassium by medical indication
* do not consume any type of salt for medical indication
* known primary or secondary hyperaldosteronism
* known severe kidney disease (routine biochemical measurement of kidney function will not be performed in household members not included in the study).
* Pregnancy or lactation
* Evidence of hyperkalemia and/or a creatinine clearance (calculated through the CKD-EPI formula <30 ml/min/1.73m2) in baseline blood laboratory. For those participants who consent to be tested, blood sample will be used. For those participant who has a laboratory test performed with those biomarkers in the past 6 months those results will be considered
* Households in which any of the study participants consume more than 50% of their meals prepared outside their home will also be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2490 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-04-14 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure at day 120 | 120 days
  Systolic Blood Pressure will be measured by a standardized automated device

SECONDARY OUTCOMES:
Hyperkalemia | 120 days
  Evidence of Hyperkalemia is determined by clinical suspicion or biochemical value defined as a serum potassium value above 5.5 mmol/l (in case it is measured) during the follow up.
Salt substitutes acceptance and incorporation into the diet | 120 days
  Salt substitutes acceptance and incorporation into the diet will be measured through a questionnaire administrated at 30 days and follow-up.
  The questionnaire includes the following questions: How many days in the last week did you use study salt? If you were meant to use the study salt in the last week but did not use it every day, what is the reason? If you use the study salt in the last week: How did you use it? How many meals did you use the study salt during the day? Did you enjoy the taste? (1 = disliked a lot; 10 = liked a lot)
Diastolic Blood Pressure at day 120 | 120 days
  Diastolic Blood Pressure will be measured by a standardized automated device
Mean arterial pressure (MAP) at day 120 | 120 days
  Systolic and Diastolic Blood Pressure will be measured by a standardized automated device in order to compute MAP

CONTACTS AND LOCATIONS:
Overall Officials: María Luz Diaz, MD, Principal Investigator — ECLA- Estudios Clínicos Latino América
Locations (1):
- IIC-Instituto de Investigaciones Clínicas, Rosario, Santa Fe Province, Argentina